CLINICAL TRIAL: NCT04266132
Title: Ultrasound Guided Retrolaminar Block Versus Ilioinguinal Nerve Block for Surgery of Inguinal Hernia in Children
Brief Title: Ultrasound Guided Retrolaminar Block for Pediatric Inguinal Hernia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahmoud Mohammed Alseoudy (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Mohammed Alseoudy, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.20.01.718
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Inguinal Hernia; Pediatric
Keywords: Retrolaminar block; Ilioinguinal nerve block
MeSH Terms: conditions — Hernia, Inguinal | interventions — Anesthesia, General; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)The study subjects and the resident assessing the outcomes will be blinded to the study group. A single investigator will assess the patients for eligibility, obtain written informed consent, open the sealed opaque envelopes containing group allocation, perform the block, and administer bupivacaine solution.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrolamianar block (RLB) (Active Comparator): General anaesthesia will be induced.Ultrasound-guided RLB will be performed under strict aseptic precautions with patient in the lateral position.The anesthetic solution will be injected.
  Interventions: Procedure: General anaesthesia; Procedure: Ultrasound-guided RLB; Drug: Bupivacaine
- Ilioinguinal nerve block (INB) (Active Comparator): General anaesthesia will be induced. Ultrasound-guided INB will be performed under strict aseptic precautions with patient in the supine position.The anesthetic solution will be injected.
  Interventions: Procedure: General anaesthesia; Procedure: Ultrasound-guided INB; Drug: Bupivacaine

INTERVENTIONS:
Procedure: General anaesthesia — General anaesthesia will be induced with 8% sevoflurane in oxygen and maintained with 1 MAC sevoflurane via a laryngeal mask.
Procedure: Ultrasound-guided RLB — The suggested ultrasound transducer orientation is sagittal paramedian (cephalacaudad direction). We begin our ultrasound scanning in a paramedian sagittal plane by finding desired level (T12- L1).The transverse process view, the costotransverse ligament can be visualized above the paravertebral space. Continuing to scan from lateral to medial, the vertebral laminae come into view.
  Arms: Retrolamianar block (RLB)
Procedure: Ultrasound-guided INB — A high-frequency probe is placed medial to the anterior superior iliac spine with the axis facing the umbilicus. A needle is inserted toward the ilioinguinal nerve as it runs between the transversus abdominis and internal oblique.
  Arms: Ilioinguinal nerve block (INB)
Drug: Bupivacaine — 0.3 ml.kg of 0.25% bupivacaine will be injected under visualization.

SUMMARY:
Regional analgesia for inguinal hernia repair in children has attracted increasing interest and different techniques like Caudal block, lumbar epidural block, wound infiltration, Ilio-inguinal nerve block and paravertebral block have been used with varying success. Ilio-inguinal nerve blockade has been widely used in this context but the duration of the block is also limited to the early postoperative period. Paravertebral blockade has been shown to produce long lasting postoperative analgesia when used in combination with general anaesthesia in paediatric herniorrhaphy . Ultrasound-guided retrolaminar block is one of the newer and technically simpler alternatives to the traditional PV block . The aim of this study is to test the efficacy and safety of ultrasound guided retrolaminar block(RLB) as an analgesic technique in surgery of pediatric inguinal hernia in comparison with with ilioinguinal nerve block(INB). It is hypothesized that RLB block will provide longer duration of postoperative analgesia than INB with few side effects.

DETAILED DESCRIPTION:
Regional analgesia for inguinal hernia repair in children has attracted increasing interest over the past few years. Caudal block, lumbar epidural block and wound infiltration using a variety of local anesthetic drugs and adjuncts have been used with varying success. Ilio-inguinal nerve blockade has been widely used in this context and despite being generally safe, complications may occurr. The duration of ilio-inguinal nerve block is also limited to the early postoperative period. Paravertebral blockade has been shown to produce long lasting postoperative analgesia when used in combination with general anaesthesia in paediatric herniorrhaphy, and has also been proposed as an alternative to general anaesthesia in adult inguinal hernia repair. Ultrasound-guided retrolaminar block is one of the newer and technically simpler alternatives to the traditional PV block. The first case report of a landmark lamina technique was followed by a study in mastectomy patients where this "blind" technique was used to inject local anesthetic between the thoracic laminae and the deep paraspinous muscles. This technique would logically decrease the chances of pleural injury, while the risk of inadvertent neuraxial injection remains. ultrasound guidance has improved the lamina technique, defining the site of injection as "retrolaminar" by real-time sonographic identification of the lamina and the needle tip-lamina contact, thus minimizing the risk of epidural injection associated with the blind technique. This was immediately followed by a report by the same group describing their first experiences with the retrolaminar technique in patients with multiple rib fractures.To our knowledge, no studies have demonstrated the efficacy and safety of ultrasound guided retro-laminar block in pediatric patients. Therefore, this study will be conducted to evaluate the efficacy and safety of retrolaminar block and compare it with the ilioinguinal nerve block in pediatric patients undergoing unilateral inguinal hernia repair. The study will include 60 patients who will be scheduled for elective outpatient inguinal herniorrhaphy. Patients will be randomly allocated using computer generated random numbers to one of two treatment groups: ultrasound guided ilio-inguinal nerve block (INB Group, n =30) or ultrasound guided retrolaminar block (RLB Group, n =30) using the sealed opaque envelope technique. The eligible patients for this study will be preoperatively evaluated regarding their medical history, clinical examination, laboratory results (complete blood picture, coagulation profile). The day before the surgery, the study protocol will be explained to parents of all patients in the study who will be kept fasting prior to surgery. General anaesthesia will be induced with 8% sevoflurane in oxygen via a facemask. After establishing venous access, a laryngeal mask will be placed and anaesthesia was maintained with 1 MAC sevoflurane and oxygen. Intraoperative monitoring included ECG, heart rate, pulse oximetry, non-invasive blood pressure and end tidal carbon dioxide concentration.During the operation, any haemodynamic changes in excess of 15% from baseline values resulted in a step-wise increase or decrease of the sevoflurane concentration. 0.3 ml.kg of 0.25% bupivacaine will be injected at the level of L1 lamina in RLB group. 0.3 ml.kg of 0.25% bupivacaine will be injected between the transversus abdominis and internal oblique toward the ilioinguinal nerve in INB group. Systolic blood pressure and heart rate will be recorded immediately prior to skin incision (baseline), 60 s after skin incision, during sac traction and on closure of the wound. Pain levels will be assessed post operatively using FLACC (face, legs, activity, cry, consolability) scale at 30 minutes and at 1, 2, 4, 6, 12, 24 hours by trained nurses and second anesthesist who will be blinded to group allocation. When the FLACC score is more than 2 and less than or equal to 5, 15 mg/kg acetaminophen IV will be administered. When the FLACC score is more than 5, 0.5μg/kg fentanyl IV will be coadministered with acetaminophen in the recovery room. Parents will be informed about the pain evaluation, and when patients have pain at home, parents will give 7 mg/kg oral ibuprofen. The anesthesiologist will record data received from the parents over the phone. Parental satisfaction after surgery will be recorded. Satisfaction levels of the parents will be given verbally as a level from 1 to 10, with the lowest level of satisfaction at a value of 1 and the highest level at 10.

ELIGIBILITY:
Inclusion Criteria:

* • American Society of Anesthesiologists (ASA) status: 1 or 2 .

  * Unilateral inguinal hernia

Exclusion Criteria:

* •spinal abnormality

  * bilateral inguinal hernia repair
  * Bleeding or coagulation diathesis.
  * History of known sensitivity to the used anesthetics.
  * Parental refusal of consent.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-05-17 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-11-20 (Estimated)

PRIMARY OUTCOMES:
First analgesic request | [Time Frame: Up to 24 hours after the procedure]
  The time of the first analgesic request will be recorded.

SECONDARY OUTCOMES:
Improvement in pain score | [Time Frame: Up to 24 hours after the procedure]
  Pain levels will be assessed post operatively using FLACC (face, legs, activity, cry, consolability) scale at 30 minutes and at 1, 2, 4, 6, 12, 24 hours
Levels of parental satisfaction after surgery | .[Time Frame: Up to 24hours after the procedure]
  Satisfaction levels of the parents will be given verbally as a level from 1 to 10, with the lowest level of satisfaction at a value of 1 and the highest level at 10
Incidence of adverse effects | [Time Frame: Up to 24 hours after the procedure]
  nausea, vomiting, hematoma, or allergic reactions will be recorded
Changes in heart rate | [Time Frame: Up to 24 hours after the procedure]
  heart rate will be recorded immediately prior to skin incision (baseline), 60 s after skin incision, during sac traction and on closure of the wound
Changes in systolic blood pressure | [Time Frame: Up to 24 hours after the procedure]
  Systolic blood pressure will be recorded immediately prior to skin incision (baseline), 60 s after skin incision, during sac traction and on closure of the wound

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Alseoudy, MD, Principal Investigator — Faculty of Medicine, Mansoura University
Locations (1):
- Mansoura university children hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No